CLINICAL TRIAL: NCT02018861
Title: A Phase 1/2, Open-Label, Dose Escalation, Safety and Tolerability Study of INCB050465 and Iitacitinib in Subjects With Previously Treated B-Cell Malignancies (CITADEL-101)
Brief Title: A Phase 1/2, Open-Label, Dose Escalation, Safety and Tolerability Study of INCB050465 and Itacitinib in Subjects With Previously Treated B-Cell Malignancies (CITADEL-101)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: INCB 50465-101 (CITADEL-101); Parsaclisib (Other: Incyte Corporation)
Record Dates: First submitted 2013-12-05; First posted 2013-12-23 (Estimated); Results first posted 2022-06-28 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: B-Cell Malignancies
MeSH Terms: interventions — parsaclisib; itacitinib; INCB039110; Rituximab; Ifosfamide; Carboplatin; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

ARMS (10):
- Parsaclisib 5 mg QD (Experimental): Parsaclisib 5 milligrams (mg) as an oral tablet once a day (QD) in 21-day treatment cycles
  Interventions: Drug: Parsaclisib
- Parsaclisib 10 mg QD (Experimental): Parsaclisib 10 mg as oral tablets QD in 21-day treatment cycles
  Interventions: Drug: Parsaclisib
- Parsaclisib 15 mg QD (Experimental): Parsaclisib 15 mg as oral tablets QD in 21-day treatment cycles
  Interventions: Drug: Parsaclisib
- Parsaclisib 20 mg QD (Experimental): Parsaclisib 15 mg as oral tablets QD in 21-day treatment cycles
  Interventions: Drug: Parsaclisib
- Parsaclisib 30 mg QD (Experimental): Parsaclisib 30 mg as oral tablets QD in 21-day treatment cycles
  Interventions: Drug: Parsaclisib
- Parsaclisib 45 mg QD (Experimental): Parsaclisib 45 mg as oral tablets QD in 21-day treatment cycles
  Interventions: Drug: Parsaclisib
- Parsaclisib 20 mg + itacitinib (INCB039110) 300 mg (Experimental): Parsaclisib 20 mg as oral tablets QD and itacitinib (INCB039110) 300 mg as oral tablets QD in 21-day treatment cycles
  Interventions: Drug: Parsaclisib; Drug: Itacitinib
- Parsaclisib 30 mg + itacitinib (INCB039110) 300 mg (Experimental): Parsaclisib 30 mg as oral tablets QD and itacitinib (INCB039110) 300 mg as oral tablets QD in 21-day treatment cycles
  Interventions: Drug: Parsaclisib; Drug: Itacitinib
- Parsaclisib 15 mg QD + R-ICE (Placebo Comparator): Parsaclisib 15 mg as oral tablets QD in 21-day treatment cycles. R-ICE was a standard-of-care chemotherapy combination administered at the following doses: rituximab 375 milligrams per meters squared (mg/m^2) intravenously (IV) on Day 1 and Day 2 of Cycle 1 and on Day 1 of Cycles 2 and 3, ifosfamide 5000 mg/m^2 IV on Day 3 of each cycle, carboplatin area under the curve (AUC) = 5 (maximum dose 800 mg) IV on Day 3 of each cycle, and etoposide 100 mg/m^2 or at doses consistent with institutional practice with approval from the medical monitor on Days 3 and 5 of each cycle. Each cycle was 21 days in duration
  Interventions: Drug: Parsaclisib; Drug: Rituximab; Drug: Ifosfamide; Drug: Carboplatin; Drug: Etoposide
- Parsaclisib 20 mg QD + R-ICE (Placebo Comparator): 20 mg as oral tablets QD in 21-day treatment cycles. R-ICE was a standard-of-care chemotherapy combination administered at the following doses: rituximab 375 mg/m^2 IV on Day 1 and Day 2 of Cycle 1 and on Day 1 of Cycles 2 and 3, ifosfamide 5000 mg/m^2 IV on Day 3 of each cycle, carboplatin AUC = 5 (maximum dose 800 mg) IV on Day 3 of each cycle, and etoposide 100 mg/m^2 or at doses consistent with institutional practice with approval from the medical monitor on Days 3 and 5 of each cycle. Each cycle was 21 days in duration.
  Interventions: Drug: Parsaclisib; Drug: Rituximab; Drug: Ifosfamide; Drug: Carboplatin; Drug: Etoposide

INTERVENTIONS:
Drug: Parsaclisib
  Other Names: INCB050465
Drug: Itacitinib
  Other Names: INCB039110; itacitinib (INCB039110)
  Arms: Parsaclisib 20 mg + itacitinib (INCB039110) 300 mg; Parsaclisib 30 mg + itacitinib (INCB039110) 300 mg
Drug: Rituximab
  Arms: Parsaclisib 15 mg QD + R-ICE; Parsaclisib 20 mg QD + R-ICE
Drug: Ifosfamide
  Arms: Parsaclisib 15 mg QD + R-ICE; Parsaclisib 20 mg QD + R-ICE
Drug: Carboplatin
  Arms: Parsaclisib 15 mg QD + R-ICE; Parsaclisib 20 mg QD + R-ICE
Drug: Etoposide
  Arms: Parsaclisib 15 mg QD + R-ICE; Parsaclisib 20 mg QD + R-ICE

SUMMARY:
Open-label, dose-escalation study in subjects with previously treated B-cell malignancies to find maximum tolerated dose (MTD) or pharmacologic active dose of a PI3Kδ inhibitor, parsaclisib, as monotherapy and in combination with: itacitinib (INCB039110), a JAK1 inhibitor; rituximab; and rituximab, ifosfamide, carboplatin, and etoposide. Parsaclisib inhibits PI3Kδ, a protein involved in growth and survival of B-cell cancer cells.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older, with lymphoid malignancies of B-cell origin including:

  1. Indolent / aggressive B-cell non-Hodgkin's lymphoma (NHL)

     * EXCLUDING: Burkitt's lymphoma and precursor B lymphoblastic leukemia/lymphoma
     * INCLUDING: any non-Hodgkin's B cell malignancy such as chronic lymphocytic leukemia (CLL) and rare non-Hodgkin's B- cell subtypes such as hairy cell leukemia, Waldenström macroglobulinemia (WM), mantle cell leukemia (MCL), and transformed NHL histologies
  2. Hodgkin's lymphoma (HL)
* Life expectancy of 12 weeks or longer
* Subject must have received ≥ 1 prior treatment regimen(s)
* The subject must not be a candidate for potentially curative therapy including hematopoietic stem cell transplantation, except where one of the standard therapy regimen combinations may be used prior to transplantation per standard medical practice

Exclusion Criteria:

* Has history of brain metastasis, spinal cord compression (unless treated, asymptomatic, and stable on most recent imaging and enrolling in expansion cohort), or lymphoma involving the central nervous system (CNS)
* Has an Eastern Cooperative Oncology Group (ECOG) performance status of ≥ 3 (≥ 2 during dose escalation)
* Received allogeneic hematopoietic stem cell transplant within the last 6 months, or has active graft versus host disease (GVHD) following allogeneic transplant, or currently receiving immunosuppressive therapy following allogeneic transplant
* Received autologous hematopoietic stem cell transplant within the last 3 months
* Inadequate marrow reserve assessed by hematologic laboratory parameters
* Inadequate renal or liver function
* Known HIV infection, or hepatitis B virus (HBV) or hepatitis C virus (HCV) viremia or at risk for HBV reactivation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2016-09-22 (Actual); Primary Completion 2021-04-12 (Actual); Study Completion 2021-04-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Corrado, M.D., Study Director — Incyte Corporation
Locations (7):
- United States (7):
  - University of Alabama At Birmingham Comprehensive Cancer Center, Birmingham, Alabama
  - University of Michigan Cancer Center, Ann Arbor, Michigan
  - Karmanos Cancer Institute, Detroit, Michigan
  - Nyu Langone Laura and Isaac Perlmutter Cancer Center, New York, New York
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - Greenville Health System Cancer Institute, Greenville, South Carolina
  - Baylor Charles A. Sammons Cancer Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Forero-Torres A, Ramchandren R, Yacoub A, Wertheim MS, Edenfield WJ, Caimi P, Gutierrez M, Akard L, Escobar C, Call J, Persky D, Iyer S, DeMarini DJ, Zhou L, Chen X, Dawkins F, Phillips TJ. Parsaclisib, a potent and highly selective PI3Kdelta inhibitor, in patients with relapsed or refractory B-cell malignancies. Blood. 2019 Apr 18;133(16):1742-1752. doi: 10.1182/blood-2018-08-867499. Epub 2019 Feb 25. PMID 30803990
- See also: Plain Language Summary of Results — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217471&parentIdentifier=INCB%2050465-101%20(CITADEL-101)&attachmentIdentifier=6ddb7eec-3da9-4cb3-9314-d18fba66dcf1&fileName=INCB50465-101_Plain_Language_Summary.pdf&versionIdentifier=b51ae8b4-81b4-46d5-ac8f-4efa98145f43

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 13 study centers in the United States.
Pre-assignment Details: This was a 4-part study. Part 1 parsaclisib monotherapy dose escalation determined the recommended dose(s) (RDs) to explore. Part 2 evaluated the combination of parsaclisib and itacitinib to determine the RDs. Part 3 expansion further evaluated the RDs of parsaclisib as monotherapy and in combination with itacitinib in disease cohorts. Part 6 consisted of a safety assessment of parsaclisib in combination with the chemotherapy regimen R-ICE (rituximab, ifosfamide, carboplatin, and etoposide).
Groups:
- Parsaclisib 5 mg QD: Participants self-administered parsaclisib 5 milligrams (mg) as an oral tablet once a day (QD) in 21-day treatment cycles.
- Parsaclisib 10 mg QD: Participants self-administered parsaclisib 10 mg as oral tablets QD in 21-day treatment cycles.
- Parsaclisib 15 mg QD: Participants self-administered parsaclisib 15 mg as oral tablets QD in 21-day treatment cycles.
- Parsaclisib 20 mg QD: Participants self-administered parsaclisib 20 mg as oral tablets QD in 21-day treatment cycles.
- Parsaclisib 30 mg QD: Participants self-administered parsaclisib 30 mg as oral tablets QD in 21-day treatment cycles.
- Parsaclisib 45 mg QD: Participants self-administered parsaclisib 45 mg as oral tablets QD in 21-day treatment cycles.
- Parsaclisib 20 mg + Itacitinib 300 mg: Participants self-administered parsaclisib 20 mg as oral tablets QD and itacitinib 300 mg as oral tablets QD in 21-day treatment cycles.
- Parsaclisib 30 mg + Itacitinib 300 mg: Participants self-administered parsaclisib 30 mg as oral tablets QD and itacitinib 300 mg as oral tablets QD in 21-day treatment cycles.
- Parsaclisib 15 mg QD + R-ICE: Participants self-administered parsaclisib 15 mg as oral tablets QD in 21-day treatment cycles. R-ICE was a standard-of-care chemotherapy combination administered at the following doses: rituximab 375 milligrams per meters squared (mg/m^2) intravenously (IV) on Day 1 and Day 2 of Cycle 1 and on Day 1 of Cycles 2 and 3, ifosfamide 5000 mg/m^2 IV on Day 3 of each cycle, carboplatin area under the curve (AUC) = 5 (maximum dose 800 mg) IV on Day 3 of each cycle, and etoposide 100 mg/m^2 or at doses consistent with institutional practice with approval from the medical monitor on Days 3 and 5 of each cycle. Each cycle was 21 days in duration.
- Parsaclisib 20 mg QD + R-ICE: Participants self-administered parsaclisib 20 mg as oral tablets QD in 21-day treatment cycles. R-ICE was a standard-of-care chemotherapy combination administered at the following doses: rituximab 375 mg/m^2 IV on Day 1 and Day 2 of Cycle 1 and on Day 1 of Cycles 2 and 3, ifosfamide 5000 mg/m^2 IV on Day 3 of each cycle, carboplatin AUC = 5 (maximum dose 800 mg) IV on Day 3 of each cycle, and etoposide 100 mg/m^2 or at doses consistent with institutional practice with approval from the medical monitor on Days 3 and 5 of each cycle. Each cycle was 21 days in duration.
Period: Parsaclisib Monotherapy: 21-day Cycles
Arm/Group | Parsaclisib 5 mg QD | Parsaclisib 10 mg QD | Parsaclisib 15 mg QD | Parsaclisib 20 mg QD | Parsaclisib 30 mg QD | Parsaclisib 45 mg QD | Parsaclisib 20 mg + Itacitinib 300 mg | Parsaclisib 30 mg + Itacitinib 300 mg | Parsaclisib 15 mg QD + R-ICE | Parsaclisib 20 mg QD + R-ICE
Started | 1 | 3 | 3 | 34 | 27 | 4 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 1 | 3 | 3 | 30 | 27 | 4 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 2 | 1 | 6 | 4 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Disease Progression | 0 | 1 | 1 | 13 | 18 | 1 | 0 | 0 | 0 | 0
Not completed — Death | 1 | 0 | 0 | 3 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Non-compliance with Study Treatment | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 4 | 1 | 2 | 0 | 0 | 0 | 0
Not completed — Unknown or Not Reported | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0
Period: Parsaclisib + Itacitinib; 21-day Cycles
Arm/Group | Parsaclisib 5 mg QD | Parsaclisib 10 mg QD | Parsaclisib 15 mg QD | Parsaclisib 20 mg QD | Parsaclisib 30 mg QD | Parsaclisib 45 mg QD | Parsaclisib 20 mg + Itacitinib 300 mg | Parsaclisib 30 mg + Itacitinib 300 mg | Parsaclisib 15 mg QD + R-ICE | Parsaclisib 20 mg QD + R-ICE
Started | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 3 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 3 | 0 | 0
Not completed — Disease Progression | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 2 | 0 | 0
Not completed — Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 0
Period: Parsaclisib + R-ICE; 21-day Cycles
Arm/Group | Parsaclisib 5 mg QD | Parsaclisib 10 mg QD | Parsaclisib 15 mg QD | Parsaclisib 20 mg QD | Parsaclisib 30 mg QD | Parsaclisib 45 mg QD | Parsaclisib 20 mg + Itacitinib 300 mg | Parsaclisib 30 mg + Itacitinib 300 mg | Parsaclisib 15 mg QD + R-ICE | Parsaclisib 20 mg QD + R-ICE
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 1
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Disease Progression | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Parsaclisib 5 mg QD | Parsaclisib 10 mg QD | Parsaclisib 15 mg QD | Parsaclisib 20 mg QD | Parsaclisib 30 mg QD | Parsaclisib 45 mg QD | Parsaclisib 20 mg + Itacitinib 300 mg | Parsaclisib 30 mg + Itacitinib 300 mg | Parsaclisib 15 mg QD + R-ICE | Parsaclisib 20 mg QD + R-ICE | Total
Number analyzed (Participants) | 1 | 3 | 3 | 34 | 27 | 4 | 8 | 3 | 4 | 1 | 88
Age, Continuous [Mean (Standard Deviation); unit: years] | NA (NA) — Due to low participant enrollment in this arm, data are not being reported, as doing so may risk participant identification. | 69.0 (16.52) | 63.3 (9.45) | 62.4 (16.48) | 63.7 (11.81) | 66.8 (8.77) | 64.6 (17.15) | 51.7 (27.02) | 62.3 (8.26) | NA (NA) — Due to low participant enrollment in this arm, data are not being reported, as doing so may risk participant identification. | 63.3 (14.44)
Sex/Gender, Customized [Number; unit: participants]
  Female | NA — Due to low participant enrollment in this arm, data are not being reported, as doing so may risk participant identification. | NA — Due to low participant enrollment in this arm, data are not being reported, as doing so may risk participant identification. | NA — Due to low participant enrollment in this arm, data are not being reported, as doing so may risk participant identification. | 12 | 14 | NA — Due to low participant enrollment in this arm, data are not being reported, as doing so may risk participant identification. | NA — Due to low participant enrollment in this arm, data are not being reported, as doing so may risk participant identification. | NA — Due to low participant enrollment in this arm, data are not being reported, as doing so may risk participant identification. | NA — Due to low participant enrollment in this arm, data are not being reported, as doing so may risk participant identification. | NA — Due to low participant enrollment in this arm, data are not being reported, as doing so may risk participant identification. | 38
  Male | NA — Due to low participant enrollment in this arm, data are not being reported, as doing so may risk participant identification. | NA — Due to low participant enrollment in this arm, data are not being reported, as doing so may risk participant identification. | NA — Due to low participant enrollment in this arm, data are not being reported, as doing so may risk participant identification. | 22 | 13 | NA — Due to low participant enrollment in this arm, data are not being reported, as doing so may risk participant identification. | NA — Due to low participant enrollment in this arm, data are not being reported, as doing so may risk participant identification. | NA — Due to low participant enrollment in this arm, data are not being reported, as doing so may risk participant identification. | NA — Due to low participant enrollment in this arm, data are not being reported, as doing so may risk participant identification. | NA — Due to low participant enrollment in this arm, data are not being reported, as doing so may risk participant identification. | 50
Race/Ethnicity, Customized [Number; unit: participants]
  Black or African American | NA — Due to low participant enrollment in this arm, data are not being reported, as doing so may risk participant identification. | NA — Due to low participant enrollment in this arm, data are not being reported, as doing so may risk participant identification. | NA — Due to low participant enrollment in this arm, data are not being reported, as doing so may risk participant identification. | 4 | 4 | NA — Due to low participant enrollment in this arm, data are not being reported, as doing so may risk participant identification. | NA — Due to low participant enrollment in this arm, data are not being reported, as doing so may risk participant identification. | NA — Due to low participant enrollment in this arm, data are not being reported, as doing so may risk participant identification. | NA — Due to low participant enrollment in this arm, data are not being reported, as doing so may risk participant identification. | NA — Due to low participant enrollment in this arm, data are not being reported, as doing so may risk participant identification. | 9
  White | NA — Due to low participant enrollment in this arm, data are not being reported, as doing so may risk participant identification. | NA — Due to low participant enrollment in this arm, data are not being reported, as doing so may risk participant identification. | NA — Due to low participant enrollment in this arm, data are not being reported, as doing so may risk participant identification. | 25 | 21 | NA — Due to low participant enrollment in this arm, data are not being reported, as doing so may risk participant identification. | NA — Due to low participant enrollment in this arm, data are not being reported, as doing so may risk participant identification. | NA — Due to low participant enrollment in this arm, data are not being reported, as doing so may risk participant identification. | NA — Due to low participant enrollment in this arm, data are not being reported, as doing so may risk participant identification. | NA — Due to low participant enrollment in this arm, data are not being reported, as doing so may risk participant identification. | 70
  Unknown or Not Reported | NA — Due to low participant enrollment in this arm, data are not being reported, as doing so may risk participant identification. | NA — Due to low participant enrollment in this arm, data are not being reported, as doing so may risk participant identification. | NA — Due to low participant enrollment in this arm, data are not being reported, as doing so may risk participant identification. | 5 | 2 | NA — Due to low participant enrollment in this arm, data are not being reported, as doing so may risk participant identification. | NA — Due to low participant enrollment in this arm, data are not being reported, as doing so may risk participant identification. | NA — Due to low participant enrollment in this arm, data are not being reported, as doing so may risk participant identification. | NA — Due to low participant enrollment in this arm, data are not being reported, as doing so may risk participant identification. | NA — Due to low participant enrollment in this arm, data are not being reported, as doing so may risk participant identification. | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: An adverse event (AE) is defined as the appearance of (or worsening of any pre-existing) undesirable sign(s), symptom(s), or medical condition(s) that occur after a participant provides informed consent. Abnormal laboratory values or test results occurring after informed consent constitute AEs only if they induce clinical signs or symptoms, are considered clinically meaningful, require therapy (e.g., hematologic abnormality that requires transfusion), or require changes in the study drug(s). A TEAE is defined as an event that was reported for the first time, or the worsening of a pre-existing event, after the first dose of study drug.
Time Frame: Up to approximately 53 months (4.4 years)
Population: Safety Population: all participants enrolled in the study who received at least 1 dose of parsaclisib, itacitinib, rituximab, ifosfamide, carboplatin, and/or etoposide
Measure: Count of Participants; unit: Participants
Arm/Group | Parsaclisib 5 mg QD | Parsaclisib 10 mg QD | Parsaclisib 15 mg QD | Parsaclisib 20 mg QD | Parsaclisib 30 mg QD | Parsaclisib 45 mg QD | Parsaclisib 20 mg + Itacitinib 300 mg | Parsaclisib 30 mg + Itacitinib 300 mg | Parsaclisib 15 mg QD + R-ICE | Parsaclisib 20 mg QD + R-ICE
Number analyzed (Participants) | 1 | 3 | 3 | 34 | 27 | 4 | 8 | 3 | 4 | 1
Participants | 1 | 3 | 3 | 32 | 25 | 4 | 6 | 3 | 4 | 1

2. Secondary Outcome: Part 1: Overall Response Rate (Percentage of Participants With Complete Response [CR] and Partial Response [PR]) Based on International Workshop on Chronic Lymphocytic Leukemia (IWCLL) Criteria for Chronic Lymphocytic Leukemia (CLL) for CLL Participants
Description: CR: (a) peripheral blood lymphocytes <4 x 10^9/Liter (L); (b) no significant lymphadenopathy and lymph nodes <1.5 centimeters (cm) in longest diameter; (c) no splenomegaly/hepatomegaly; (d) no disease-related constitutional symptoms; (e) neutrophils ≥1.5 x 10^9/L; (f) platelets ≥100 x 10^9/L; (g) hemoglobin ≥11.0 grams/deciliter (g/dL) (without transfusion); (h) minimal residual disease assessment; (i) normocellular marrow, with no CLL cells/no B-lymphoid nodules. PR (improvement in ≥2 Group A parameters and ≥1 Group B parameter if previously abnormal. If only 1 parameter of both Groups A and B was abnormal before therapy, only 1 needs to improve): Group A: (a) decrease of ≥50% (from Baseline) in lymph nodes, liver/spleen size, and circulating lymphocyte count; (b) any constitutional symptoms. Group B: (a) platelets ≥100 x 10^9/L or increase ≥50% over Baseline; (b) hemoglobin ≥11 g/dL or increase ≥50% over Baseline; (c) presence of CLL cells or B-lymphoid nodules.
Time Frame: Up to approximately 53 months (4.4 years)
Population: Intent-to-Treat (ITT) Population: all participants with CLL enrolled in the study who received at least 1 dose of parsaclisib, itacitinib, rituximab, ifosfamide, carboplatin, and/or etoposide. Confidence intervals were calculated based on the exact method for binomial distributions.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Parsaclisib 5 mg QD | Parsaclisib 10 mg QD | Parsaclisib 15 mg QD | Parsaclisib 20 mg QD | Parsaclisib 30 mg QD | Parsaclisib 45 mg QD
Number analyzed (Participants) | 0 | 1 | 0 | 1 | 3 | 1
percentage of participants |  | 0.0 [0.0 to 97.5] |  | 0.0 [0.0 to 97.5] | 66.7 [9.4 to 99.2] | 0.0 [0.0 to 97.5]

3. Secondary Outcome: Part 2: Overall Response Rate (Percentage of Participants With CR and PR) Based on IWCLL Criteria for CLL for Participants With CLL
Description: CR: (a) peripheral blood lymphocytes <4 x 10^9/L; (b) no significant lymphadenopathy and lymph nodes <1.5 cm in longest diameter; (c) no splenomegaly/hepatomegaly; (d) no disease-related constitutional symptoms; (e) neutrophils ≥1.5 x 10^9/L; (f) platelets ≥100 x 10^9/L; (g) hemoglobin ≥11.0 g/dL (without transfusion); (h) minimal residual disease assessment; (i) normocellular marrow, with no CLL cells/no B-lymphoid nodules. PR (improvement in ≥2 Group A parameters and ≥1 Group B parameter if previously abnormal. If only 1 parameter of both Groups A and B was abnormal before therapy, only 1 needs to improve): Group A: (a) decrease of ≥50% (from Baseline) in lymph nodes, liver/spleen size, and circulating lymphocyte count; (b) any constitutional symptoms. Group B: (a) platelets ≥100 x 10^9/L or increase ≥50% over Baseline; (b) ≥11 g/dL or increase ≥50% over Baseline; (c) presence of CLL cells or B-lymphoid nodules.
Time Frame: Up to approximately 44 months (3.7 years)
Population: ITT Population: all participants with CLL. Confidence intervals were calculated based on the exact method for binomial distributions.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Parsaclisib 20 mg + Itacitinib 300 mg | Parsaclisib 30 mg + Itacitinib 300 mg
Number analyzed (Participants) | 1 | 0
percentage of participants | 100.0 [2.5 to 100.0] |

4. Secondary Outcome: Part 6: Overall Response Rate (Percentage of Participants With CR and PR) Based on IWCLL Criteria for CLL for Participants With CLL
Description: as for outcome 3
Time Frame: Up to approximately 4 months
Population: ITT Population: all participants with CLL
Arm/Group | Parsaclisib 15 mg QD + R-ICE | Parsaclisib 20 mg QD + R-ICE
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Part 1: ORR Based on the VIth International Workshop on Waldenström Macroglobulinemia (WM) Response Assessment for Participants With WM
Description: ORR: sum of participants achieving minor response (MR), PR, very good partial response (VGPR), and CR. CR: (a) no serum monoclonal IgM protein by immunofixation; (b) normal serum IgM level; (c) complete resolution of extramedullary disease, i.e., lymphadenopathy/splenomegaly if present at Baseline (BL); (d) morphologically normal bone marrow aspirate and trephine biopsy. VGPR: (a) detectable monoclonal IgM protein; (b) ≥90% reduction in serum IgM level from BL; (c) complete resolution of extramedullary disease, i.e., lymphadenopathy/splenomegaly if present at BL; (d) no new signs/symptoms of active disease. PR: (a) detectable monoclonal IgM protein; (b) ≥50% but <90% reduction in serum IgM level from BL; (c) reduction in extramedullary disease, i.e., lymphadenopathy/splenomegaly if present at BL; (d) no new signs/symptoms of active disease. MR: (a) detectable monoclonal IgM protein; (b) ≥25% but <50% reduction in serum IgM level from BL; (d) no new signs/symptoms of active disease.
Time Frame: Up to approximately 53 months (4.4 years)
Population: ITT Population: all participants with WM. Confidence intervals were calculated based on the exact method for binomial distributions.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Parsaclisib 5 mg QD | Parsaclisib 10 mg QD | Parsaclisib 15 mg QD | Parsaclisib 20 mg QD | Parsaclisib 30 mg QD | Parsaclisib 45 mg QD
Number analyzed (Participants) | 0 | 0 | 0 | 1 | 0 | 0
percentage of participants |  |  |  | 100.0 [2.5 to 100.0] |  |

6. Secondary Outcome: Part 2: ORR Based on the VIth International Workshop on WM Response Assessment for Participants With WM
Description: ORR: sum of participants achieving MR, PR, VGPR, and CR. CR: (a) no serum monoclonal IgM protein by immunofixation; (b) normal serum IgM level; (c) complete resolution of extramedullary disease, i.e., lymphadenopathy/splenomegaly if present at BL; (d) morphologically normal bone marrow aspirate and trephine biopsy. VGPR: (a) detectable monoclonal IgM protein; (b) ≥90% reduction in serum IgM level from BL; (c) complete resolution of extramedullary disease, i.e., lymphadenopathy/splenomegaly if present at BL; (d) no new signs/symptoms of active disease. PR: (a) detectable monoclonal IgM protein; (b) ≥50% but <90% reduction in serum IgM level from BL; (c) reduction in extramedullary disease, i.e., lymphadenopathy/splenomegaly if present at BL; (d) no new signs/symptoms of active disease. MR: (a) detectable monoclonal IgM protein; (b) ≥25% but <50% reduction in serum IgM level from BL; (d) no new signs/symptoms of active disease.
Time Frame: Up to approximately 44 months (3.7 years)
Population: as for outcome 5
Arm/Group | Parsaclisib 20 mg + Itacitinib 300 mg | Parsaclisib 30 mg + Itacitinib 300 mg
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Part 6: ORR Based on the VIth International Workshop on WM Response Assessment for Participants With WM
Description: as for outcome 6
Time Frame: Up to approximately 4 months
Population: ITT Population: all participants with WM
Arm/Group | Parsaclisib 15 mg QD + R-ICE | Parsaclisib 20 mg QD + R-ICE
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Part 1: ORR (Sum of Participants With CR and PR) Based on the Revised Response Criteria for Hodgkin's Lymphoma (HL) and Non-Hodgkin's Lymphoma (NHL), Using Positron Emission Tomography-computed Tomography (PET-CT) and CT
Description: CR, PET-CT: (a) complete metabolic response (MR); (b) lymph nodes and extralymphatic sites (LNs/ELSs): score 1, 2, or 3, with/without residual mass; (c) no new lesions (NNLs); (d) no evidence of fluorodeoxyglucose-avid disease in marrow. CT: complete radiologic response: (a) regression of target nodes/nodal masses to ≤ 1.5 cm in longest transverse lesion diameter; (b) no ELSs of disease; (c) absence of nonmeasured lesions; (d) regression to normal organ size; (e) NNLs; (f) normal morphological bone marrow. PR, PET-CT: (a) partial MR; (b) LNs/ELSs: score 4 or 5, with reduced uptake compared with Baseline and residual mass of any size; (c) NNLs; (d) residual uptake higher than uptake in normal marrow but reduced compared with Baseline. CT: partial remission: (a) LNs/ELSs: ≥ 50% decrease in the sum of the product of the perpendicular diameters for multiple lesions of up to 6 target measurable sites; (b) spleen must have regressed by > 50% in length beyond normal; (c) NNLs.
Time Frame: Up to approximately 53 months (4.4 years)
Population: ITT Population: all participants with the indicated types of HL and NHL. Confidence intervals were calculated based on the exact method for binomial distributions.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Parsaclisib 5 mg QD | Parsaclisib 10 mg QD | Parsaclisib 15 mg QD | Parsaclisib 20 mg QD | Parsaclisib 30 mg QD | Parsaclisib 45 mg QD
Number analyzed (Participants) | 1 | 2 | 3 | 32 | 24 | 3
percentage of participants
  Diffuse large B-cell lymphoma: number analyzed (Participants) | 1 | 1 | 2 | 11 | 6 | 2
  Diffuse large B-cell lymphoma | 0.0 [0.0 to 97.5] | 0.0 [0.0 to 97.5] | 50.0 [1.3 to 98.7] | 36.4 [10.9 to 69.2] | 16.7 [0.4 to 64.1] | 50.0 [1.3 to 98.7]
  Follicular lymphoma: number analyzed (Participants) | 0 | 1 | 1 | 7 | 5 | 0
  Follicular lymphoma |  | 100.0 [2.5 to 100.0] | 100.0 [2.5 to 100.0] | 85.7 [42.1 to 99.6] | 40.0 [5.3 to 85.3] |
  Mantle cell lymphoma: number analyzed (Participants) | 0 | 0 | 0 | 6 | 2 | 1
  Mantle cell lymphoma |  |  |  | 66.7 [22.3 to 95.7] | 100.0 [15.8 to 100.0] | 0.0 [0.0 to 97.5]
  Marginal zone lymphoma: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0
  Marginal zone lymphoma |  |  |  |  | 0.0 [0.0 to 97.5] |
  Extranodal marginal zone lymphoma of mucosa-associated lymphatic tissue: number analyzed (Participants) | 0 | 0 | 0 | 2 | 0 | 0
  Extranodal marginal zone lymphoma of mucosa-associated lymphatic tissue |  |  |  | 50.0 [1.3 to 98.7] |  |
  Nodal marginal zone B-cell lymphoma: number analyzed (Participants) | 0 | 0 | 0 | 1 | 3 | 0
  Nodal marginal zone B-cell lymphoma |  |  |  | 100.0 [2.5 to 100.0] | 100.0 [29.2 to 100.0] |
  Splenic marginal zone lymphoma: number analyzed (Participants) | 0 | 0 | 0 | 1 | 1 | 0
  Splenic marginal zone lymphoma |  |  |  | 100.0 [2.5 to 100.0] | 100.0 [2.5 to 100.0] |
  Classical Hodgkin's lymphoma: number analyzed (Participants) | 0 | 0 | 0 | 4 | 5 | 0
  Classical Hodgkin's lymphoma |  |  |  | 50.0 [6.8 to 93.2] | 0.0 [0.0 to 52.2] |
  Nodular lymphocytic-predominant Hodgkin's lymphoma: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0
  Nodular lymphocytic-predominant Hodgkin's lymphoma |  |  |  |  | 0.0 [0.0 to 97.5] |

9. Secondary Outcome: Part 2: ORR (Sum of Participants With CR and PR) Based on the Revised Response Criteria for HL and NHL, Using PET-CT and CT
Description: CR, PET-CT: (a) complete MR; (b) LNs/ELSs: score 1, 2, or 3, with/without residual mass; (c) NNLs; (d) no evidence of fluorodeoxyglucose-avid disease in marrow. CT: complete radiologic response: (a) regression of target nodes/nodal masses to ≤ 1.5 cm in longest transverse lesion diameter; (b) no ELSs of disease; (c) absence of nonmeasured lesions; (d) regression to normal organ size; (e) NNLs; (f) normal morphological bone marrow. PR, PET-CT: (a) partial MR; (b) LNs/ELSs: score 4 or 5, with reduced uptake compared with Baseline and residual mass of any size; (c) NNLs; (d) residual uptake higher than uptake in normal marrow but reduced compared with Baseline. CT: partial remission: (a) LNs/ELSs: ≥ 50% decrease in the sum of the product of the perpendicular diameters for multiple lesions of up to 6 target measurable sites; (b) spleen must have regressed by > 50% in length beyond normal; (c) NNLs.
Time Frame: Up to approximately 44 months (3.7 years)
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Parsaclisib 20 mg + Itacitinib 300 mg | Parsaclisib 30 mg + Itacitinib 300 mg
Number analyzed (Participants) | 7 | 3
percentage of participants
  Diffuse large B-cell lymphoma: number analyzed (Participants) | 3 | 3
  Diffuse large B-cell lymphoma | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8]
  Follicular lymphoma: number analyzed (Participants) | 1 | 0
  Follicular lymphoma | 0.0 [0.0 to 97.5] |
  Mantle cell lymphoma: number analyzed (Participants) | 1 | 0
  Mantle cell lymphoma | 100.0 [2.5 to 100.0] |
  Marginal zone lymphoma: number analyzed (Participants) | 0 | 0
  Extranodal marginal zone lymphoma of mucosa-associated lymphatic tissue: number analyzed (Participants) | 0 | 0
  Nodal marginal zone B-cell lymphoma: number analyzed (Participants) | 0 | 0
  Splenic marginal zone lymphoma: number analyzed (Participants) | 0 | 0
  Classical Hodgkin's lymphoma: number analyzed (Participants) | 2 | 0
  Classical Hodgkin's lymphoma | 50.0 [1.3 to 98.7] |
  Nodular lymphocytic-predominant Hodgkin's lymphoma: number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Part 6: ORR (Sum of Participants With CR and PR) Based on the Revised Response Criteria for HL and NHL, Using PET-CT and CT
Description: as for outcome 9
Time Frame: Up to approximately 4 months
Population: ITT Population: all participants with the indicated types of HL and NHL
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Parsaclisib 15 mg QD + R-ICE | Parsaclisib 20 mg QD + R-ICE
Number analyzed (Participants) | 4 | 1
percentage of participants
  Diffuse large B-cell lymphoma | 50.0 [NA to NA] — Summary statistics are not available due to the small sample size in Part 6. | 100.0 [NA to NA] — Summary statistics are not available due to the small sample size in Part 6.
  Follicular lymphoma: number analyzed (Participants) | 0 | 0
  Mantle cell lymphoma: number analyzed (Participants) | 0 | 0
  Marginal zone lymphoma: number analyzed (Participants) | 0 | 0
  Extranodal marginal zone lymphoma of mucosa-associated lymphatic tissue: number analyzed (Participants) | 0 | 0
  Nodal marginal zone B-cell lymphoma: number analyzed (Participants) | 0 | 0
  Splenic marginal zone lymphoma: number analyzed (Participants) | 0 | 0
  Classical Hodgkin's lymphoma: number analyzed (Participants) | 0 | 0
  Nodular lymphocytic-predominant Hodgkin's lymphoma: number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Cmax of Itacitinib in Combination With Parsaclisib
Description: Cmax is defined as the maximum observed plasma or serum concentration of itacitinib.
Time Frame: Cycle 1 Day 15; pre-dose and 0.5, 1, 2, 4, 6, 8, and 12 hours post-dose
Population: Pharmacokinetic (PK)/Pharmacodynamics (PD) Population: participants in the ITT/Safety Population who had PK/PD data. Data from the parsaclisib 20 mg + itacitinib 300 mg and the parsaclisib 30 mg + itacitinib 300 mg arms were pooled for analysis because all participants received 300 mg itacitinib and there is no drug-drug interaction between parsaclisib and itacitinib to affect the PK of either drug.
Measure: Mean (Standard Deviation); unit: nanomoles (nmol)
Groups:
- Parsaclisib 20/30 mg + Itacitinib 300 mg: Participants self-administered parsaclisib 20 mg or 30 mg as oral tablets QD and itacitinib 300 mg as oral tablets QD in 21-day treatment cycles.
Arm/Group | Parsaclisib 20/30 mg + Itacitinib 300 mg
Number analyzed (Participants) | 7
nanomoles (nmol) | 887 (404)

12. Secondary Outcome: Tmax of Itacitinib in Combination With Parsaclisib
Description: tmax is defined as the time to the maximum concentration of itacitinib.
Time Frame: Cycle 1 Day 15; pre-dose and 0.5, 1, 2, 4, 6, 8, and 12 hours post-dose
Population: PK/PD Population. Data from the parsaclisib 20 mg + itacitinib 300 mg and the parsaclisib 30 mg + itacitinib 300 mg arms were pooled for analysis because all participants received 300 mg itacitinib and there is no drug-drug interaction between parsaclisib and itacitinib to affect the PK of either drug.
Measure: Median (Full Range); unit: hours
Groups:
- Parsaclisib 20/30 mg + Itacitinib 300 mg: Participants self-administered parsaclisib 20 or 30 mg as oral tablets QD and itacitinib 300 mg as oral tablets QD in 21-day treatment cycles.
Arm/Group | Parsaclisib 20/30 mg + Itacitinib 300 mg
Number analyzed (Participants) | 7
hours | 2.0 [1.0 to 4.0]

13. Secondary Outcome: Cmin of Itacitinib in Combination With Parsaclisib
Description: Cmin is defined as the minimum observed plasma or serum concentration over the dose interval of itacitinib.
Time Frame: Cycle 1 Day 15; pre-dose and 0.5, 1, 2, 4, 6, 8, and 12 hours post-dose
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: nmol
Arm/Group | Parsaclisib 20/30 mg + Itacitinib 300 mg
Number analyzed (Participants) | 7
nmol | 32.8 (32.5)

14. Secondary Outcome: AUC0-t of Itacitinib in Combination With Parsaclisib
Description: AUC0-t is defined as the area under the plasma or serum concentration-time curve from time = 0 to the last measurable concentration at time = t of itacitinib.
Time Frame: Cycle 1 Day 15; pre-dose and 0.5, 1, 2, 4, 6, 8, and 12 hours post-dose
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: hours (hr)*nmol/L
Arm/Group | Parsaclisib 20/30 mg + Itacitinib 300 mg
Number analyzed (Participants) | 7
hours (hr)*nmol/L | 6450 (3780)

15. Secondary Outcome: AUC0-τ of Itacitinib in Combination With Parsaclisib
Description: AUC0-τ is defined as the area under the steady-state plasma or serum concentration-time curve over 1 dose interval (i.e., from hour 0 to 12 for once every 12 hours [q12h] administration or from hour 0 to 24 for once every 24 hours [q24h] administration) of itacitinib.
Time Frame: Cycle 1 Day 15; pre-dose and 0.5, 1, 2, 4, 6, 8, and 12 hours post-dose
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: hr*nmol/L
Arm/Group | Parsaclisib 20/30 mg + Itacitinib 300 mg
Number analyzed (Participants) | 7
hr*nmol/L | 6450 (13780)

16. Secondary Outcome: Parts 1 and 2: Cmax of Parsaclisib as Monotherapy and in Combination With Itacitinib
Description: Cmax is defined as the maximum observed plasma or serum concentration of parsaclisib. PK samples collected in Part 2, the combination dose escalation study, and in Part 3, Cohort E expansion group, were analyzed for both parsaclisib and itacitinib.
Time Frame: Cycle 1 Days 1 and 15; pre-dose and 0.5, 1, 2, 4, 6, 8, and 12 hours post-dose
Population: PK/PD Population. Only participants with available data were analyzed. In the combination therapy arms, data are reported for the Part 3 Cohort E population (participants with B-cell malignancies).
Measure: Mean (Standard Deviation); unit: nmol
Arm/Group | Parsaclisib 5 mg QD | Parsaclisib 10 mg QD | Parsaclisib 15 mg QD | Parsaclisib 20 mg QD | Parsaclisib 30 mg QD | Parsaclisib 45 mg QD | Parsaclisib 20 mg + Itacitinib 300 mg | Parsaclisib 30 mg + Itacitinib 300 mg
Number analyzed (Participants) | 1 | 3 | 3 | 4 | 4 | 4 | 8 | 3
nmol
  Cycle 1 Day 1 | 354 (NA) — Standard deviation was not calculated for a single participant. | 791 (502) | 808 (316) | 1270 (655) | 3270 (775) | 4010 (1400) | 1740 (1010) | 2040 (338)
  Cycle 1 Day 15: number analyzed (Participants) | 1 | 3 | 3 | 4 | 3 | 4 | 8 | 3
  Cycle 1 Day 15 | 690 (NA) — Standard deviation was not calculated for a single participant. | 856 (449) | 1310 (290) | 1280 (437) | 3310 (682) | 5530 (3210) | 2390 (1480) | 2500 (973)

17. Secondary Outcome: Parts 1 and 2: Tmax of Parsaclisib as Monotherapy and in Combination With Itacitinib
Description: tmax is defined as the time to the maximum concentration of parsaclisib. PK samples collected in Part 2, the combination dose escalation study, and in Part 3, Cohort E expansion group, were analyzed for both parsaclisib and itacitinib.
Time Frame: Cycle 1 Days 1 and 15; pre-dose and 0.5, 1, 2, 4, 6, 8, and 12 hours post-dose
Population: as for outcome 16
Measure: Median (Full Range); unit: hours
Arm/Group | Parsaclisib 5 mg QD | Parsaclisib 10 mg QD | Parsaclisib 15 mg QD | Parsaclisib 20 mg QD | Parsaclisib 30 mg QD | Parsaclisib 45 mg QD | Parsaclisib 20 mg + Itacitinib 300 mg | Parsaclisib 30 mg + Itacitinib 300 mg
Number analyzed (Participants) | 1 | 3 | 3 | 4 | 4 | 4 | 8 | 3
hours
  Cycle 1 Day 1 | 2.0 [2.0 to 2.0] | 1.0 [0.5 to 2.0] | 1.0 [1.0 to 2.0] | 1.0 [0.5 to 2.0] | 0.5 [0.5 to 1.0] | 1.0 [0.5 to 2.0] | 1.0 [0.5 to 1.0] | 1.0 [1.0 to 1.0]
  Cycle 1 Day 15: number analyzed (Participants) | 1 | 3 | 3 | 4 | 3 | 4 | 8 | 3
  Cycle 1 Day 15 | 0.5 [0.5 to 0.5] | 1.0 [0.5 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [0.5 to 1.0] | 0.5 [0.5 to 2.0] | 0.5 [0.5 to 1.0] | 1.0 [0.5 to 2.0] | 1.0 [0.5 to 1.0]

18. Secondary Outcome: Parts 1 and 2: Cmin of Parsaclisib as Monotherapy and in Combination With Itacitinib
Description: Cmin is defined as the minimum observed plasma or serum concentration over the dose interval of parsaclisib. PK samples collected in Part 2, the combination dose escalation study, and in Part 3, Cohort E expansion group, were analyzed for both parsaclisib and itacitinib.
Time Frame: Cycle 1 Days 1 and 15; pre-dose and 0.5, 1, 2, 4, 6, 8, and 12 hours post-dose
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: nmol
Arm/Group | Parsaclisib 5 mg QD | Parsaclisib 10 mg QD | Parsaclisib 15 mg QD | Parsaclisib 20 mg QD | Parsaclisib 30 mg QD | Parsaclisib 45 mg QD | Parsaclisib 20 mg + Itacitinib 300 mg | Parsaclisib 30 mg + Itacitinib 300 mg
Number analyzed (Participants) | 1 | 3 | 3 | 4 | 4 | 4 | 8 | 3
nmol
  Cycle 1 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Cycle 1 Day 15: number analyzed (Participants) | 1 | 3 | 3 | 4 | 3 | 4 | 8 | 3
  Cycle 1 Day 15 | 127 (NA) — Standard deviation was not calculated for a single participant. | 104 (46) | 156 (99.8) | 178 (141) | 295 (83.1) | 864 (690) | 515 (652) | 341 (278)

19. Secondary Outcome: Parts 1 and 2: AUC0-t of Parsaclisib as Monotherapy and in Combination With Itacitinib
Description: AUC0-t is defined as the area under the plasma or serum concentration-time curve from time = 0 to the last measurable concentration at time = t of parsaclisib. PK samples collected in Part 2, the combination dose escalation study, and in Part 3, Cohort E expansion group, were analyzed for both parsaclisib and itacitinib.
Time Frame: Cycle 1 Days 1 and 15; pre-dose and 0.5, 1, 2, 4, 6, 8, and 12 hours post-dose
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: hr*nmol/L
Arm/Group | Parsaclisib 5 mg QD | Parsaclisib 10 mg QD | Parsaclisib 15 mg QD | Parsaclisib 20 mg QD | Parsaclisib 30 mg QD | Parsaclisib 45 mg QD | Parsaclisib 20 mg + Itacitinib 300 mg | Parsaclisib 30 mg + Itacitinib 300 mg
Number analyzed (Participants) | 1 | 3 | 3 | 4 | 4 | 4 | 8 | 3
hr*nmol/L
  Cycle 1 Day 1 | 2110 (NA) — Standard deviation was not calculated for a single participant. | 3260 (1460) | 3730 (678) | 5990 (2650) | 13300 (2480) | 16800 (4880) | 7540 (3370) | 10400 (1330)
  Cycle 1 Day 15: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

20. Secondary Outcome: Parts 1 and 2: AUC0-τ of Parsaclisib as Monotherapy and in Combination With Itacitinib
Description: AUC0-τ is defined as the area under the steady-state plasma or serum concentration-time curve over 1 dose interval (i.e., from hour 0 to 12 for q12h administration or from hour 0 to 24 for q24h administration) of parsaclisib. PK samples collected in Part 2, the combination dose escalation study, and in Part 3, Cohort E expansion group, were analyzed for both parsaclisib and itacitinib.
Time Frame: Cycle 1 Days 1 and 15; pre-dose and 0.5, 1, 2, 4, 6, 8, and 12 hours post-dose
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: hr*nmol/L
Arm/Group | Parsaclisib 5 mg QD | Parsaclisib 10 mg QD | Parsaclisib 15 mg QD | Parsaclisib 20 mg QD | Parsaclisib 30 mg QD | Parsaclisib 45 mg QD | Parsaclisib 20 mg + Itacitinib 300 mg | Parsaclisib 30 mg + Itacitinib 300 mg
Number analyzed (Participants) | 1 | 3 | 3 | 4 | 4 | 4 | 8 | 3
hr*nmol/L
  Cycle 1 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Cycle 1 Day 15 | 7130 (NA) — Standard deviation was not calculated for a single participant. | 6910 (2330) | 11100 (6310) | 11900 (5110) | 24800 (2140) | 47700 (30500) | 22400 (17100) | 22900 (10700)

21. Secondary Outcome: Part 3: Cmax of Parsaclisib Monotherapy
Description: Cmax is defined as the maximum observed plasma or serum concentration of parsaclisib. PK samples for parsaclisib monotherapy were collected and analyzed from the Part 3 dose expansion (different participant populations). Cohort A: B-cell malignancies; Cohort B: Hodgkin's lymphoma; Cohort C: diffuse large B-cell lymphoma; Cohort D: indolent lymphoma.
Time Frame: Cycle 1 Days 1 and 15; pre-dose and 0.5, 1, 2, 4, 6, 8, and 12 hours post-dose
Population: PK/PD Population. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: nmol
Arm/Group | Parsaclisib 5 mg QD | Parsaclisib 10 mg QD | Parsaclisib 15 mg QD | Parsaclisib 20 mg QD | Parsaclisib 30 mg QD | Parsaclisib 45 mg QD
Number analyzed (Participants) | 0 | 0 | 0 | 30 | 23 | 0
nmol
  Cycle 1 Day 1, Cohort A: number analyzed (Participants) | 0 | 0 | 0 | 17 | 8 | 0
  Cycle 1 Day 1, Cohort A |  |  |  | 1550 (544) | 2350 (944) |
  Cycle 1 Day 15, Cohort A: number analyzed (Participants) | 0 | 0 | 0 | 15 | 9 | 0
  Cycle 1 Day 15, Cohort A |  |  |  | 1720 (492) | 2390 (648) |
  Cycle 1 Day 1, Cohort B: number analyzed (Participants) | 0 | 0 | 0 | 1 | 6 | 0
  Cycle 1 Day 1, Cohort B |  |  |  | 1200 (NA) — Standard deviation was not calculated for a single participant. | 1720 (925) |
  Cycle 1 Day 15, Cohort B: number analyzed (Participants) | 0 | 0 | 0 | 1 | 6 | 0
  Cycle 1 Day 15, Cohort B |  |  |  | 1930 (NA) — Standard deviation was not calculated for a single participant. | 2260 (784) |
  Cycle 1 Day 1, Cohort C: number analyzed (Participants) | 0 | 0 | 0 | 9 | 4 | 0
  Cycle 1 Day 1, Cohort C |  |  |  | 1760 (772) | 1760 (534) |
  Cycle 1 Day 15, Cohort C: number analyzed (Participants) | 0 | 0 | 0 | 8 | 4 | 0
  Cycle 1 Day 15, Cohort C |  |  |  | 2060 (682) | 3920 (1320) |
  Cycle 1 Day 1, Cohort D: number analyzed (Participants) | 0 | 0 | 0 | 3 | 4 | 0
  Cycle 1 Day 1, Cohort D |  |  |  | 1760 (580) | 2500 (279) |
  Cycle 1 Day 15, Cohort D: number analyzed (Participants) | 0 | 0 | 0 | 3 | 4 | 0
  Cycle 1 Day 15, Cohort D |  |  |  | 1600 (378) | 2990 (783) |

22. Secondary Outcome: Part 3: Tmax of Parsaclisib Monotherapy
Description: tmax is defined as the time to the maximum concentration of parsaclisib. PK samples for parsaclisib monotherapy were collected and analyzed from the Part 3 dose expansion (different participant populations). Cohort A: B-cell malignancies; Cohort B: Hodgkin's lymphoma; Cohort C: diffuse large B-cell lymphoma; Cohort D: indolent lymphoma.
Time Frame: Cycle 1 Days 1 and 15; pre-dose and 0.5, 1, 2, 4, 6, 8, and 12 hours post-dose
Population: PK/PD Population. Only participants with available data were analyzed.
Measure: Median (Full Range); unit: hours
Arm/Group | Parsaclisib 5 mg QD | Parsaclisib 10 mg QD | Parsaclisib 15 mg QD | Parsaclisib 20 mg QD | Parsaclisib 30 mg QD | Parsaclisib 45 mg QD
Number analyzed (Participants) | 0 | 0 | 0 | 30 | 23 | 0
hours
  Cycle 1 Day 1, Cohort A: number analyzed (Participants) | 0 | 0 | 0 | 17 | 8 | 0
  Cycle 1 Day 1, Cohort A |  |  |  | 0.5 [0.5 to 4.0] | 1.0 [0.5 to 2.0] |
  Cycle 1 Day 15, Cohort A: number analyzed (Participants) | 0 | 0 | 0 | 15 | 9 | 0
  Cycle 1 Day 15, Cohort A |  |  |  | 1.0 [0.5 to 1.0] | 1.0 [0.5 to 2.0] |
  Cycle 1 Day 1, Cohort B: number analyzed (Participants) | 0 | 0 | 0 | 1 | 6 | 0
  Cycle 1 Day 1, Cohort B |  |  |  | 2.0 [2.0 to 2.0] | 1.5 [0.5 to 2.0] |
  Cycle 1 Day 15, Cohort B: number analyzed (Participants) | 0 | 0 | 0 | 1 | 6 | 0
  Cycle 1 Day 15, Cohort B |  |  |  | 0.5 [0.5 to 0.5] | 0.75 [0.5 to 8.0] |
  Cycle 1 Day 1, Cohort C: number analyzed (Participants) | 0 | 0 | 0 | 9 | 4 | 0
  Cycle 1 Day 1, Cohort C |  |  |  | 0.5 [0.5 to 4.0] | 1.0 [0.5 to 2.0] |
  Cycle 1 Day 15, Cohort C: number analyzed (Participants) | 0 | 0 | 0 | 8 | 4 | 0
  Cycle 1 Day 15, Cohort C |  |  |  | 1.0 [0.5 to 1.0] | 0.5 [0.5 to 0.5] |
  Cycle 1 Day 1, Cohort D: number analyzed (Participants) | 0 | 0 | 0 | 3 | 4 | 0
  Cycle 1 Day 1, Cohort D |  |  |  | 1.0 [0.5 to 1.0] | 0.75 [0.5 to 1.0] |
  Cycle 1 Day 15, Cohort D: number analyzed (Participants) | 0 | 0 | 0 | 3 | 4 | 0
  Cycle 1 Day 15, Cohort D |  |  |  | 0.5 [0.5 to 1.0] | 1.0 [0.5 to 1.0] |

23. Secondary Outcome: Part 3: Cmin of Parsaclisib Monotherapy
Description: Cmin is defined as the minimum observed plasma or serum concentration over the dose interval of parsaclisib. PK samples for parsaclisib monotherapy were collected and analyzed from the Part 3 dose expansion (different participant populations). Cohort A: B-cell malignancies; Cohort B: Hodgkin's lymphoma; Cohort C: diffuse large B-cell lymphoma; Cohort D: indolent lymphoma.
Time Frame: Cycle 1 Days 1 and 15; pre-dose and 0.5, 1, 2, 4, 6, 8, and 12 hours post-dose
Population: PK/PD Population. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: nmol
Arm/Group | Parsaclisib 5 mg QD | Parsaclisib 10 mg QD | Parsaclisib 15 mg QD | Parsaclisib 20 mg QD | Parsaclisib 30 mg QD | Parsaclisib 45 mg QD
Number analyzed (Participants) | 0 | 0 | 0 | 30 | 23 | 0
nmol
  Cycle 1 Day 1, Cohort A: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0
  Cycle 1 Day 15, Cohort A: number analyzed (Participants) | 0 | 0 | 0 | 15 | 9 | 0
  Cycle 1 Day 15, Cohort A |  |  |  | 214 (171) | 281 (137) |
  Cycle 1 Day 1, Cohort B: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0
  Cycle 1 Day 15, Cohort B: number analyzed (Participants) | 0 | 0 | 0 | 1 | 6 | 0
  Cycle 1 Day 15, Cohort B |  |  |  | 395 (NA) — Standard deviation was not calculated for a single participant. | 296 (177) |
  Cycle 1 Day 1, Cohort C: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0
  Cycle 1 Day 15, Cohort C: number analyzed (Participants) | 0 | 0 | 0 | 8 | 4 | 0
  Cycle 1 Day 15, Cohort C |  |  |  | 197 (79.6) | 477 (137) |
  Cycle 1 Day 1, Cohort D: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0
  Cycle 1 Day 15, Cohort D: number analyzed (Participants) | 0 | 0 | 0 | 3 | 4 | 0
  Cycle 1 Day 15, Cohort D |  |  |  | 202 (161) | 421 (365) |

24. Secondary Outcome: Part 3: AUC0-t of Parsaclisib Monotherapy
Description: AUC0-t is defined as the area under the plasma or serum concentration-time curve from time = 0 to the last measurable concentration at time = t of of parsaclisib. PK samples for parsaclisib monotherapy were collected and analyzed from the Part 3 dose expansion (different participant populations). Cohort A: B-cell malignancies; Cohort B: Hodgkin's lymphoma; Cohort C: diffuse large B-cell lymphoma; Cohort D: indolent lymphoma.
Time Frame: Cycle 1 Days 1 and 15; pre-dose and 0.5, 1, 2, 4, 6, 8, and 12 hours post-dose
Population: PK/PD Population. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: hr*nmol/L
Arm/Group | Parsaclisib 5 mg QD | Parsaclisib 10 mg QD | Parsaclisib 15 mg QD | Parsaclisib 20 mg QD | Parsaclisib 30 mg QD | Parsaclisib 45 mg QD
Number analyzed (Participants) | 0 | 0 | 0 | 30 | 23 | 0
hr*nmol/L
  Cycle 1 Day 1, Cohort A: number analyzed (Participants) | 0 | 0 | 0 | 17 | 8 | 0
  Cycle 1 Day 1, Cohort A |  |  |  | 6530 (2280) | 10700 (4150) |
  Cycle 1 Day 15, Cohort A: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0
  Cycle 1 Day 1, Cohort B: number analyzed (Participants) | 0 | 0 | 0 | 1 | 6 | 0
  Cycle 1 Day 1, Cohort B |  |  |  | 7010 (NA) — Standard deviation was not calculated for a single participant. | 8430 (3560) |
  Cycle 1 Day 15, Cohort B: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0
  Cycle 1 Day 1, Cohort C: number analyzed (Participants) | 0 | 0 | 0 | 9 | 4 | 0
  Cycle 1 Day 1, Cohort C |  |  |  | 7110 (2760) | 12000 (3230) |
  Cycle 1 Day 15, Cohort C: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0
  Cycle 1 Day 1, Cohort D: number analyzed (Participants) | 0 | 0 | 0 | 3 | 4 | 0
  Cycle 1 Day 1, Cohort D |  |  |  | 7230 (2530) | 9970 (1260) |
  Cycle 1 Day 15, Cohort D: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

25. Secondary Outcome: Part 3: AUC0-τ of Parsaclisib Monotherapy
Description: AUC0-τ is defined as the area under the steady-state plasma or serum concentration-time curve over 1 dose interval (i.e., from hour 0 to 12 for once every 12 hours [q12h] administration or from hour 0 to 24 for once every 24 hours [q24h] administration) of parsaclisib. PK samples for parsaclisib monotherapy were collected and analyzed from the Part 3 dose expansion (different participant populations). Cohort A: B-cell malignancies; Cohort B: Hodgkin's lymphoma; Cohort C: diffuse large B-cell lymphoma; Cohort D: indolent lymphoma.
Time Frame: Cycle 1 Days 1 and 15; pre-dose and 0.5, 1, 2, 4, 6, 8, and 12 hours post-dose
Population: PK/PD Population. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: hr*nmol/L
Arm/Group | Parsaclisib 5 mg QD | Parsaclisib 10 mg QD | Parsaclisib 15 mg QD | Parsaclisib 20 mg QD | Parsaclisib 30 mg QD | Parsaclisib 45 mg QD
Number analyzed (Participants) | 0 | 0 | 0 | 30 | 23 | 0
hr*nmol/L
  Cycle 1 Day 1, Cohort A: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0
  Cycle 1 Day 15, Cohort A: number analyzed (Participants) | 0 | 0 | 0 | 15 | 9 | 0
  Cycle 1 Day 15, Cohort A |  |  |  | 12600 (5170) | 19500 (6020) |
  Cycle 1 Day 1, Cohort B: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0
  Cycle 1 Day 15, Cohort B: number analyzed (Participants) | 0 | 0 | 0 | 1 | 6 | 0
  Cycle 1 Day 15, Cohort B |  |  |  | 17900 (NA) — Standard deviation was not calculated for a single participant. | 20100 (6640) |
  Cycle 1 Day 1, Cohort C: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0
  Cycle 1 Day 15, Cohort C: number analyzed (Participants) | 0 | 0 | 0 | 8 | 4 | 0
  Cycle 1 Day 15, Cohort C |  |  |  | 14200 (4600) | 28000 (4310) |
  Cycle 1 Day 1, Cohort D: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0
  Cycle 1 Day 15, Cohort D: number analyzed (Participants) | 0 | 0 | 0 | 3 | 4 | 0
  Cycle 1 Day 15, Cohort D |  |  |  | 13600 (7270) | 25200 (8820) |

ADVERSE EVENTS:
Time Frame: Up to approximately 53 months (4.4 years)
Description: Treatment-emergent adverse events (TEAEs), defined as events that were reported for the first time, or the worsening of a pre-existing event, after the first dose of study drug, are reported for the Safety Population, defined as all participants enrolled in the study who received at least 1 dose of parsaclisib, itacitinib, rituximab, ifosfamide, carboplatin, and/or etoposide.
Groups:
- Total: All participants in all treatment arms combined.
Arm/Group | Parsaclisib 5 mg QD | Parsaclisib 10 mg QD | Parsaclisib 15 mg QD | Parsaclisib 20 mg QD | Parsaclisib 30 mg QD | Parsaclisib 45 mg QD | Parsaclisib 20 mg + Itacitinib 300 mg | Parsaclisib 30 mg + Itacitinib 300 mg | Parsaclisib 15 mg QD + R-ICE | Parsaclisib 20 mg QD + R-ICE | Total
All-Cause Mortality (participants affected / at risk) | 1/1 | 0/3 | 0/3 | 3/34 | 1/27 | 0/4 | 0/8 | 0/3 | 0/4 | 0/1 | 5/88
Serious Adverse Events (participants affected / at risk) | 1/1 | 2/3 | 1/3 | 14/34 | 12/27 | 2/4 | 0/8 | 2/3 | 1/4 | 1/1 | 36/88
Other Adverse Events (participants affected / at risk) | 1/1 | 3/3 | 3/3 | 32/34 | 24/27 | 4/4 | 6/8 | 3/3 | 4/4 | 1/1 | 81/88
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Parsaclisib 5 mg QD (N=1) | Parsaclisib 10 mg QD (N=3) | Parsaclisib 15 mg QD (N=3) | Parsaclisib 20 mg QD (N=34) | Parsaclisib 30 mg QD (N=27) | Parsaclisib 45 mg QD (N=4) | Parsaclisib 20 mg + Itacitinib 300 mg (N=8) | Parsaclisib 30 mg + Itacitinib 300 mg (N=3) | Parsaclisib 15 mg QD + R-ICE (N=4) | Parsaclisib 20 mg QD + R-ICE (N=1) | Total (N=88)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anal incontinence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (2)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (5)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cytomegalovirus colitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Dermatitis exfoliative (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (6)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Escherichia bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastritis erosive (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 2 (3)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Klebsiella bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Renal tubular necrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
White blood cell count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Parsaclisib 5 mg QD (N=1) | Parsaclisib 10 mg QD (N=3) | Parsaclisib 15 mg QD (N=3) | Parsaclisib 20 mg QD (N=34) | Parsaclisib 30 mg QD (N=27) | Parsaclisib 45 mg QD (N=4) | Parsaclisib 20 mg + Itacitinib 300 mg (N=8) | Parsaclisib 30 mg + Itacitinib 300 mg (N=3) | Parsaclisib 15 mg QD + R-ICE (N=4) | Parsaclisib 20 mg QD + R-ICE (N=1) | Total (N=88)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (6) | 6 (6) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 12 (13)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Abdominal tenderness (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 8 (9)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 5 (5)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 5 (8) | 4 (5) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 15 (19)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 5 (5)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 6 (6) | 6 (8) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 16 (18)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 6 (11) | 3 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 10 (16)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 5 (5)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 7 (7) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 11 (11)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 6 (6) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 9 (9)
Blood cholesterol increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 4 (7)
Blood phosphorus increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Candida infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (5)
Cerumen impaction (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (6) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 10 (11)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 9 (9) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 16 (16)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (2) | 5 (5) | 11 (13) | 0 (0) | 4 (5) | 0 (0) | 1 (1) | 0 (0) | 23 (27)
Deafness (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 8 (8) | 4 (4) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 16 (16)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (7)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 14 (19) | 11 (16) | 1 (1) | 2 (3) | 1 (1) | 1 (1) | 0 (0) | 31 (42)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2) | 6 (7) | 7 (8) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 17 (21)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 8 (8)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (2) | 3 (3) | 4 (4) | 0 (0) | 1 (2) | 0 (0) | 1 (2) | 0 (0) | 11 (14)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (6)
Eye irritation (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (6)
Fatigue (General disorders) | 0 (0) | 1 (1) | 1 (1) | 11 (12) | 9 (9) | 1 (1) | 5 (6) | 1 (1) | 1 (1) | 0 (0) | 30 (32)
Fluid overload (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 2 (4)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Genital discomfort (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 6 (7) | 0 (0) | 1 (3) | 0 (0) | 2 (2) | 0 (0) | 11 (14)
Hepatic steatosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 5 (5)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (14) | 3 (3) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 10 (20)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 2 (5) | 1 (1) | 1 (2) | 0 (0) | 9 (13)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 6 (8) | 4 (5) | 0 (0) | 1 (1) | 0 (0) | 2 (7) | 0 (0) | 15 (23)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 4 (6)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 4 (4) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 6 (10)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 5 (5) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 9 (9)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 5 (5)
Lacrimation increased (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (2)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Middle ear inflammation (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (4) | 1 (1) | 4 (4) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 10 (13)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (2)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (5)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 2 (2) | 1 (1) | 1 (4) | 0 (0) | 1 (1) | 0 (0) | 10 (13)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2) | 9 (10) | 12 (15) | 1 (1) | 3 (3) | 2 (2) | 1 (1) | 0 (0) | 32 (36)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 7 (7)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 5 (5)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 7 (10) | 7 (16) | 1 (1) | 1 (2) | 0 (0) | 3 (6) | 1 (1) | 20 (36)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 4 (5)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 6 (7) | 3 (3) | 2 (2) | 1 (2) | 0 (0) | 1 (1) | 1 (1) | 15 (17)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 0 (0) | 5 (5) | 4 (4) | 0 (0) | 1 (2) | 0 (0) | 1 (2) | 0 (0) | 12 (14)
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 2 (4)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (5)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 4 (5)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 7 (9)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 4 (4)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (5)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 7 (7)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Polycythaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 8 (9) | 3 (6) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 13 (17)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 2 (2) | 0 (0) | 6 (8) | 2 (5) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 12 (17)
Radiculopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 1 (1) | 8 (10) | 2 (2) | 2 (2) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 17 (20)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Renal impairment (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory syncytial virus test positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (5)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 6 (7)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spinal cord compression (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 7 (7)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 4 (5) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 9 (10)
Taste disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 7 (12) | 5 (6) | 0 (0) | 0 (0) | 0 (0) | 3 (9) | 1 (2) | 17 (30)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 2 (3)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Transaminases increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2) | 1 (3) | 3 (4) | 4 (4) | 1 (1) | 3 (7) | 0 (0) | 0 (0) | 0 (0) | 14 (21)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 2 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (10)
Vaginal discharge (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Visual perseveration (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 1 (3)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 4 (4) | 11 (11) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 1 (1) | 21 (22)
Weight decreased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (5)
Weight increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 5 (7)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 3 (8) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 7 (12)
White blood cell count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Wound infection bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Wound infection pseudomonas (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Following the first publication, the Institution and/or Principal Investigator may publish data or results from the Study, provided, however, that the Institution and/or Principal Investigator submits the proposed publication to the Sponsor for review at least sixty (60) days prior to the date of the proposed publication. Sponsor may remove from the proposed publication any information that is considered confidential and/or proprietary other than Study data and results.

DOCUMENTS (2):
  • Study Protocol (2019-08-07): https://cdn.clinicaltrials.gov/large-docs/61/NCT02018861/Prot_000.pdf
  • Statistical Analysis Plan (2015-06-26): https://cdn.clinicaltrials.gov/large-docs/61/NCT02018861/SAP_001.pdf